CLINICAL TRIAL: NCT01536652
Title: Prandial Oriented NovoMix 30® - the Physiological Insulin Therapy of Diabetes Type 2
Brief Title: Prandial Orientated Biphasic Insulin Aspart 30 Therapy - the Physiological Premix Insulin Therapy for Type 2 Diabetes
Acronym: ProMix
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1932
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Prescription at the discretion of the treating physician

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to document the glycaemic parameters, adverse events, including drug reactions, as well as hypoglycaemic episodes, in patients that switched from insulin glargine combined with oral antidiabetic drugs (OADs) to biphasic insulin aspart 30 (NovoMix® 30) combined with OADs, when applicable.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes mellitus type 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with diabetes mellitus type 2, using insulin glargine in combination with one or more OADs, being in inadequate glycaemic control and are indicated to receive biphasic insulin aspart 30
Sampling Method: Non-Probability Sample
Enrollment: 4994 (Actual)
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Body weight
Preprandial and postprandial blood glucose values (self measured)
Insulin dosage
Incidence of (serious) adverse drug reactions
Incidence of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com